CLINICAL TRIAL: NCT02897791
Title: Main Idea Perception of Written Stories and in Pictures Among Impaired Right Hemisphere Patients
Acronym: stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ofer Keren, MD, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-14-1529-OK-CTIL
Record Dates: First submitted 2016-07-27; First posted 2016-09-13 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Late Effects of Cerebrovascular Accident

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Impaired Rt. Hemisphere patients (Experimental): 20 first stroke patients
  Interventions: Behavioral: written evaluations
- control (Experimental): 20 healthy adults without any known damage to the right hemisphere. The two groups will be matched concerning sex, age, educational level and socio-economic status.
  Interventions: Behavioral: written evaluations

INTERVENTIONS:
Behavioral: written evaluations — answering questions about pictures and stories

SUMMARY:
Main idea perception of written stories and in pictures among impaired right hemisphere patients Abstract The right hemisphere is considered to complement the language processing abilities of the opposite hemisphere; it is responsible for the processing of secondary and unusual characteristics of linguistic stimulates. This processing enables, among other functions, the comprehension of metaphors and humor. Additionally, it enables the execution of inferring from spoken and written discourse. Studies which deal with common impairments among right-hemisphere-damaged (RHD) individuals, found that inference processing of written stories and narrative sequences presented in pictures was impaired. This impairment could damage the ability to create global coherence, which is an important component of central theme comprehension of different types of narrative. Another important component is superstructures, schemas which aid creating, remembering and producing the main ideas of spoken and written discourse. Other studies consider impairment in creating global coherence, or Theory of Mind impairment, as the source of central theme comprehension impairment among RHD individuals.

Discourse is an integral part of interpersonal communication, and of proper social conduct. The themes chosen for conversation reflect the functional role of discourse from semantic and pragmatic points of view.

The aim of the current study is to deepen the current knowledge concerning central theme comprehension among RHD individuals following cerebrovascular accident (CVA), in two genres of written discourse (classic stories and stories with a twist), and in situations represented by single pictures. Unlike written stories, the extraction of the central theme out of a single picture requires focusing on a single situation and relying on non-linguistic visual information. Differences concerning central theme comprehension in the different discourse genres and in the pictures might be able to assist in selecting diagnostic and therapeutic tools designed to work on high cognitive-linguistic abilities, which are usually impaired among RHD individuals. In later stage, these tools are meant to help improving RHD individuals' spontaneous narrative skills.

The study will include 20 RHD adults following CVA, and 20 healthy adults without any known damage to the right hemisphere. The two groups will be matched concerning sex, age, educational level and socio-economic status. The subjects will perform the study tests during three sessions, 60 minutes each. The screening tests will include language diagnosis - Western Aphasia Battery (WAB), and reading test no. 37 included in the Psycholinguistic Assessments of Language Processing in Aphasia's battery (PALPA). Patients diagnosed with aphasia will be excluded from research. The research tests will include: central theme comprehension test in stories and pictures, including classic stories, stories with a twist, and pictures of different situations (each will be accompanied by a multiple-choice question concerning the central theme), sub- exanimations taken from "Frigbi" battery designed to evaluate memory and phonological memory capacity, Raven's Progressive Colored Matrices test designed to evaluate pre-morbid abilities (non-linguistic), Theory of Mind (T.O.M) evaluation test, and tests designed to evaluate central coherence impairment: Navon Figures test for evaluation of global visual perception impairment, and Rey-Osterrieth Complex Figure Test (RCFT) - Recall Form test for evaluation of visual-perceptive organizational ability, and non-verbal memory. The performances of the two groups will be compared in each test using statistical tests. In addition, the interaction between all variables will be measured.

ELIGIBILITY:
Inclusion Criteria:

first stroke without primary diminutive impairment Hebrew as a first language

Exclusion Criteria:

previous neurological illness irritable patient

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Picture and Story Comprehension Interview Score | 1 hour
  Patients were administered the Picture and Story Comprehension Interview. This measure includes 12 short story items and 30 picture items. Regarding each item, patients were asked to choose the sentence that best represented the main idea of the picture or story (multiple choice questions). The interview score was computed as the sum of correct answers.